CLINICAL TRIAL: NCT04805177
Title: Early Minimally Invasive Image Guided Endoscopic Evacuation of Intracerebral Haemorrhage: a Prospective Pilot Study
Brief Title: Early Minimally Invasive Image Guided Endoscopic Evacuation of Intracerebral Haemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-00161, ko21Bonati
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Intracerebral Hemorrhage (ICH)
Keywords: endoscopic evacuation; pilot study; spontaneous supratentorial Intracerebral Hemorrhage (SSICH); minimally invasive image guided endoscopic surgery; early hematoma evacuation
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Intervention Model Description: single arm pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hematoma evacuation (Experimental): Early minimally invasive image guided hematoma evacuation
  Interventions: Procedure: hematoma evacuation

INTERVENTIONS:
Procedure: hematoma evacuation — early minimally invasive image guided hematoma evacuation in patients suffering from ICH

SUMMARY:
The aim of this pilot study is to provide an assessment of safety and feasibility of early minimally invasive image guided endoscopic hematoma evacuation (within 24 hours of symptom onset) in patients suffering from intracerebral haemorrhage (ICH).

DETAILED DESCRIPTION:
Spontaneous supratentorial intracerebral haemorrhage (SSICH) is the is the second most common form of stroke. The aim of this single centre, single arm pilot study is to provide an assessment of safety and feasibility of early minimally invasive image guided endoscopic hematoma evacuation (within 24 hours of symptom onset) in patients suffering from intracerebral haemorrhage (ICH).

Furthermore this study contributes to the understanding of secondary neuronal damage involved in ICH through the measurement of biomarkers for neuronal damage and their response to early hematoma evacuation.

ELIGIBILITY:
Inclusion Criteria:

* No relevant disability prior to ICH (mRS 0-1 prior to ICH)
* Primary supratentorial deep or superficial intraparenchymal ICH of volume ≥ 20 mL < 100 mL (measured using formula) demonstrated on CT or MRI, with or without a 2 component of intraventricular haemorrhage
* CT/MRI demonstrates ICH stability (< 5 mL growth) at 6 hours after the admission scan if surgery is performed >6 hours after admission CT
* NIHSS ≥ 8 OR if a patient with a NIHSS<8 presents with at least one of the following deficits:

  * a severe hemiparesis (4 motor points on the NIHSS for facial palsy, motoric upper and lower extremities combined); OR
  * a severe motor or sensory aphasia (2 points on the NIHSS); OR
  * a profound hemi-inattention (formerly neglect, 2 points on the NIHSS); OR
  * a decreased level of consciousness (GCS<13)
* Presenting GCS 5 - 15
* Endoscopic haematoma evacuation can be initiated within 24 hours of symptom onset
* Systolic blood pressure can be controlled at <160 mmHg

Exclusion Criteria:

* Imaging:

  * "Spot sign" identified on CT angiography (CTA)
  * Structural vascular or brain lesion as suspected cause of ICH, such as a vascular malformation (cavernous malformation, arteriovenous malformation (AVM) etc), aneurysm, neoplasm
  * Haemorrhagic conversion of an underlying ischemic stroke
  * Infratentorial haemorrhage
  * Large associated intra-ventricular haemorrhage requiring treatment for related mass effect or shift due to trapped ventricle (extraventricular drainage (EVD) for intracranial pressure (ICP) management is allowed)
  * Midbrain extension/involvement
* Coagulation Issues:

  * Oral or parenteral therapeutic anticoagulation which cannot be pharmacologically reverted until the planned time of evacuation
  * Known hereditary or acquired haemorrhagic diathesis, coagulation factor deficiency
  * Platelet count < 100 x 103 cells/mm3 or known platelet dysfunction
  * international normalized ratio (INR) > 1.5 for any reason, elevated prothrombin time or activated partial thromboplastin time (aPTT), which cannot be corrected or otherwise accounted for (i.e., lupus anti-coagulant)
* Presenting GCS 3 or 4
* Requirement for emergent surgical decompression or uncontrolled ICP after EVD
* Unable to obtain consent from patient or appropriate surrogate (for patients without competence)
* Pregnancy, breast-feeding, or positive pregnancy test [either serum or urine] (woman of child-bearing potential must have a negative history of current pregnancy prior to the study procedure)
* Evidence of active infection (indicated by fever ≥38°C) at the time of study inclusion
* Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 180 days
* Based on physician's judgment, patient does not have the necessary mental capacity to participate or is unwilling or unable to comply with protocol follow up appointment schedule
* Active drug or alcohol use or dependence

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-08-08 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Level of disability | 6 month after treatment onset
  level of disability 6 months after treatment, measured by the modified Rankin Scale (mRS). Good functional outcome is defined by a score on the mRS of ≤3.
Change in hematoma volume to ≤15 mL | from baseline to 24 hours after treatment
  Change in hematoma volume to ≤15 mL
number of specific adverse events (AE) | 6 month after treatment onset
  number of specific adverse events (AE) (death, ischemic stroke, recurrent ICH (defined as any increase in hematoma volume at follow-up that is associated with a worsening of the focal-neurological deficit by ≥4 points on the National Institute of Health Stroke Scale (NIHSS) and/or a decrease in consciousness by ≥2 points on the Glasgow Coma Scale (GCS), epileptic seizure, infection, any need for open neurosurgical procedures)

SECONDARY OUTCOMES:
Change in relative (percentage) hematoma volume | from baseline to 24 hours after treatment
  Change in relative (percentage) hematoma volume
Change of focal neurological deficit measured by the NIHSS | from baseline to 6 months
  Change of focal neurological deficit measured by the NIHSS. The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.
Change of serum biomarkers of brain injury | from baseline to 6 months
  Change of serum biomarkers of brain injury (light-chain neurofilament subunit (NfL), the Glial Fibrillary Acidic Protein (GFAP) and the S100 calcium-binding protein B (S100B))
Total time spent on the intensive care unit | from baseline to hospital discharge (approx. 1 month)
  Total time spent on the intensive care unit
Total time spent in intubation | from baseline to hospital discharge (approx. 1 month)
  Total time spent in intubation

CONTACTS AND LOCATIONS:
Overall Officials: Jehuda Soleman, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - Department of Neurology, University Hospital Basel, Basel
  - Department of Neurosurgery, University Hospital Basel, Basel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hallenberger TJ, Guzman R, Soleman J. Minimally invasive image-guided endoscopic evacuation of intracerebral haemorrhage: How I Do it. Acta Neurochir (Wien). 2023 Jun;165(6):1597-1602. doi: 10.1007/s00701-022-05326-3. Epub 2022 Aug 5. PMID 35930078